CLINICAL TRIAL: NCT01351415
Title: An Open-label, Randomized, Phase IIIb Trial Evaluating the Efficacy and Safety of Standard of Care +/- Continuous Bevacizumab Treatment Beyond Progression of Disease (PD) in Patients With Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC) After First Line Treatment With Bevacizumab Plus a Platinum Doublet-containing Chemotherapy
Brief Title: A Study of Bevacizumab in Combination With Standard of Care Treatment in Participants With Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22097; 2010-022645-14 (EudraCT Number)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Docetaxel; Erlotinib Hydrochloride; Pemetrexed

ARMS (2):
- Bevacizumab + Standard of Care (Experimental): Participants will receive bevacizumab on Day 1 of every 21-days cycle along with standard of care (Erlotinib or Docetaxel or Pemetrexed) as second line treatment, until the occurrence of an unacceptable toxicity or withdrawal of consent (whichever occurs first).
  Interventions: Drug: Bevacizumab; Drug: Docetaxel; Drug: Erlotinib; Drug: Pemetrexed
- Standard of Care (Active Comparator): Participants will receive investigator's choice of standard of care (Erlotinib or Docetaxel or Pemetrexed) according to local practice until the occurrence of an unacceptable toxicity or withdrawal of consent (whichever occurs first).
  Interventions: Drug: Docetaxel; Drug: Erlotinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Bevacizumab — Participants will receive bevacizumab 7.5 or 15 milligrams per kilogram (mg/kg) intravenously.
  Other Names: Avastin
  Arms: Bevacizumab + Standard of Care
Drug: Docetaxel — Docetaxel 60 or 75 milligram per meter square (mg/m^2) on Day 1 every 21 days.
Drug: Erlotinib — Erlotinib 150 mg daily taken on an empty stomach at least one hour before or two hours after the ingestion of food.
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 IV over 10 minutes on Day 1 every 21 days.

SUMMARY:
This open-label, randomized, multicenter study will evaluate the efficacy and safety of bevacizumab (Avastin) in combination with standard of care (SOC) treatment in participants with advanced non-squamous NSCLC. Participants will be enrolled at documentation of progression of disease (PD) after 4-6 cycles of first-line treatment with bevacizumab plus a platinum doublet-containing therapy and a minimum of two cycles of bevacizumab maintenance treatment prior to PD. Participants will be randomly assigned to one of two treatment arms to receive either bevacizumab plus SOC treatment or SOC treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-squamous NSCLC
* Documented progression of disease (locally recurrent or metastatic) per investigator assessment following first-line treatment with 4-6 cycles of Bevacizumab plus a platinum doublet-containing chemotherapy regimen and a minimum of 2 cycles of Bevacizumab (monotherapy) maintenance treatment prior to first progression of disease
* No treatment interruption of Bevacizumab treatment greater than 2 consecutive cycles (42 days) between the start of first-line treatment to start of Cycle 1 of second line treatment
* Randomization within 4 weeks of progression of disease
* At least one unidimensionally measurable lesion meeting RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Participants with adequate hematological, liver, and renal function
* Female participants must not be pregnant or breast-feeding. Female participants of childbearing potential and fertile male participants must agree to use a highly effective contraceptive during the trial and for a period of at least 6 months following the last administration of trial drug(s)

Exclusion Criteria:

* Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Epidermal growth factor receptor (EGFR)-mutation-positive disease according to local laboratory testing
* History of hemoptysis greater than or equal to (>/=) grade 2 within 3 months of randomization
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding and active gastrointestinal bleeding
* Major cardiac disease
* Treatment with any other investigational agent within 28 days prior to randomization
* Known hypersensitivity to bevacizumab or any of its excipients, or any SOC drugs foreseen
* Malignancy other than NSCLC within 5 years prior to randomization and evidence of any other disease that contraindicates the use of an investigational or SOC drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2011-06-25 (Actual); Primary Completion 2016-06-25 (Actual); Study Completion 2016-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (179):
- United States (68):
  - USA Mitchell Cancer Institute, Mobile, Alabama
  - Palo Verde Hema/Onc, Glendale, Arizona
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Clopton Clinic, Jonesboro, Arkansas
  - East Valley Hematology ; Oncology Medical Group, Burbank, California
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - Scripps Clinic; Hematology & Oncology, La Jolla, California
  - Sutter Cancer Center, Sacramento, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Innovative Clinical Research Institute, Whittier, California
  - The Hospital of Central CT, New Britain, Connecticut
  - Eastern Ct Hema/Onco Assoc; Dept of Oncology, Norwich, Connecticut
  - Lynn Cancer Institute - West, Boca Raton, Florida
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - Summit Cancer Care PC, Savannah, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Oncology-Evanston Nthwest Healthcare Kellogg Cancer Care Ctr, Evanston, Illinois
  - Joliet Oncology Hematology Associates, Ltd., Joliet, Illinois
  - Cancer Care & Hematology; Specialists of Chicagoland, Niles, Illinois
  - W. Suburban Ctr for Cncer Care, River Forest, Illinois
  - St. Francis Medical Group, Indianapolis, Indiana
  - Oncology Hematology Associates of Southwest Indiana, Newburgh, Indiana
  - McFarland Clinic, Ames, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Jewish Cancer Care, Louisville, Kentucky
  - Hematology/Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - York Hospital, York Village, Maine
  - Anne Arundel Health System Research Instit-Annapolis Oncology Ctr, Annapolis, Maryland
  - Tufts Medical Center; Neely Cancer Center, Boston, Massachusetts
  - Ann Arbor Hematology Oncology, Ann Arbor, Michigan
  - Henry Ford Hospital; Hematology Oncology, Detroit, Michigan
  - Cancer & Hematology Center of West Michigan, Grand Rapids, Michigan
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - St Joseph Oncology, Saint Joseph, Missouri
  - Heartland CCOP/Missouri Baptist Medical Center, St Louis, Missouri
  - Stony Brook Univ Cancer Ctr; Medical Oncology Clinic, Stony Brook, New York
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Mid Ohio Onc Hematology Inc, Columbus, Ohio
  - Dayton Clinical Oncology Prog, Dayton, Ohio
  - Signal Point Clinical; Research Center, LLC, Middletown, Ohio
  - Toledo Hospital; CCOP Toledo, Toledo, Ohio
  - Bay Area Hospital, Coos Bay, Oregon
  - St. Lukes Hospital and Health Network, Bethlehem, Pennsylvania
  - Hematology & Oncology Assoc; North Eastern Pennsylvania, Dunmore, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - University of Pennsylvania; Radiation Oncology, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - West Clinic, Germantown, Tennessee
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Unv of TX SW Med Cntr; Hematology/Onc, Dallas, Texas
  - Delta Hematology/ Oncology Associates, Portsmouth, Virginia
  - Blue Ridge Cancer Care - Roanoke, Roanoke, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Fox Valley Hema and Onc SC, Appleton, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - UNI OF WISCONSIN SCHOOL OF MEDICINE; GI Oncology Research Group, Paul P Carbone Cancer Center, Madison, Wisconsin
- Argentina (6):
  - Inst. Alexander Fleming; Oncology Dept, Buenos Aires
  - Centro Oncologico Infinito; Oncologia, La Pampa
  - Hospital Privado de Comunidad; Oncology, Mar del Plata
  - Sanatorio Parque de Rosario, Rosario
  - ISIS Clinica Especializada, Santa Fe
  - Clínica Viedma, Viedma, Rio Negro
- Austria (8):
  - LKH Hohenems; Abteilung für Pulmologie, Hohenems
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Innere Medizin Abt. Für Hämatologie & Onkologie, Innsbruck
  - Lkh Natters; Abt. Für Atemwegs- & Lungenkrankheiten, Natters
  - A.Ö. LKH; Abt. für Lungenkrankheiten, Steyr
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
  - Krankenhaus Der Stadt Wien Lainz; V. Medizinische Abt., Vienna
  - SMZ - Baumgartner Hohe, Pavilion Leopold; 1.Interne Lungenabteilung, Onkologische Tagesklinik, Vienna
  - Klinikum Wels-Grieskirchen; Lungenabt., Wels
- Clin. Europe (Ste Elisabeth), Brussels, Belgium
- Brazil (10):
  - Centro de Pesquisa Clínica- Instituto do Câncer do Ceará- ICC, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - Sociedade beneficente de senhoras Hospital Sirio Libanes, Brasília, Federal District
  - Centro de Estudos e Pesquisas Oncologicas - CESPO, Brasília, Federal District
  - Instituto de Câncer de Brasília, Taguatinga, Federal District
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- Nordsjællands Hospital, Hillerød, Onkologisk Afdeling, Hillerød, Denmark
- France (19):
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Hospitalier Intercommunal; Service de Pneumologie, Créteil
  - Hopital Nord Ouest;Unite 2c, Gleizé
  - Centre Oscar Lambret, Lille
  - Hopital Calmette; Pneumologie, Lille
  - Hopital Louis Pradel; Cardiologie B, Lyon
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - Hopital Nord; Service d'Oncologie Multidisciplinaire et Innovation Thérapeutique, Marseille
  - Centre Antoine Lacassagne, Nice
  - Ch Lyon Sud; Chir Onc Gyne Sct Jules Courmont, Pierre-Bénite
  - CH Rene Dubos; Oncologie, Pontoise
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hia Sainte Anne; Pneumologie, Toulon
  - Hopital Sainte Musse; Pneumologie, Toulon
  - Clinique Pasteur; Pneumologie, Toulouse
  - Chi De La Haute Saone De Vesoul; Pneumologie, Vesoul
- Germany (15):
  - Zentralklinik Bad Berka GmbH; Pneumologie, Bad Berka
  - Praxis Dr. med. David Borquez, Bergisch Gladbach
  - Klinikum Esslingen; Klinik für Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar
  - Krankenhaus Nordwest; Klinik f. Onkologie und Hämatologie, Frankfurt
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - LungenClinic Großhansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin I, Halle
  - Universitaetsklinikum des Saarlandes; Innere Medizin V, Homburg/Saar
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - St. Vincentius Kliniken Karlsruhe; Abteilung Hämatologie / Onkologie, Karlsruhe
  - Robert-Koch-Klinik; Pneumologie, Leipzig
  - Praxis Christian Geßner, Leipzig
  - Johannes-Wesling-Klinikum Minden; Onkologische Ambulanz / Tagesklinik, Minden
  - Ludwig-Maximilians Uni Klinik Innenstadt; Medizinische Klinik, München
  - Pius-Hospital; Klinik fuer Haematologie und Onkologie, Oldenburg
- Greece (4):
  - Sotiria Hospital, Athens
  - Metropolitan Hospital; 2Nd Oncology Clinic, Piraeus
  - General Hospital of Thessaloniki Papanikolaou; Uni Pneumonology Dept., Thessaloniki
  - Diavalkaniko Hospital, Thessaloniki
- Italy (7):
  - Citta Ospedaliera; Divisione Oncologia Medica, Avellino, Campania
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini; U.O.C. Pneumologia Ad Indirizzo Oncologico 1, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Az. Osp. Di Busto P.O. Di Saronno; U.O. Di Oncologia Medica, Saronno, Lombardy
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
- Japan (14):
  - Aichi Cancer Center Hospital; Respiratory Medicine, Aichi
  - National Cancer Center Hospital East; Thoracic Oncology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Thoracic Oncology, Ehime
  - National Hospital Organization Kyushu Cancer Center, Thoracic Oncology, Fukuoka
  - Hyogo Cancer Center; Thoracic Oncology, Hyōgo
  - Kanagawa Cardiovascular and Respiratory Center; Respiratory Medicine, Kanagawa
  - Yokohama Municipal Citizen'S Hospital; Respiratory, Kanagawa
  - Miyagi Cancer Center; Respiratory Medicine, Miyagi
  - Okayama University Hospital; Respiratory and Allergy Medicine, Okayama
  - OSAKA CITY GENERAL HOSPITAL;Medical Oncology, Osaka
  - Osaka International Cancer Institute; Thoracic Oncology, Osaka
  - Shizuoka Cancer Center; Thoracic Oncology, Shizuoka
  - National Cancer Center Hospital; Thoracic Medical Oncology, Tokyo
  - The Cancer Institute Hospital of JFCR, Respiratory Medicine, Tokyo
- Lebanon (3):
  - American University of Beirut - Medical Center, Beirut
  - Hotel Dieu de France; Oncology, Beirut
  - Middle East Inst. of Health; Oncology, Beirut
- Mexico (3):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Hospital Central Sur de Alta Especialidad Petróleos Mexicanos, Mexico City
  - Centro Médico Abc the American British Cowdray Medical Center, I.A.P. - Centro de Cáncer, Mexico City
- Netherlands (6):
  - Amphia Ziekenhuis; Afdeling Longziekten, Breda
  - Catharina Ziekenhuis; Dept of Lung Diseases, Eindhoven
  - Ziekenhuis St Jansdal; Dept of Lung Diseases, Harderwijk
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Antonius Ziekenhuis; Dept of Lung Diseases, Nieuwegein
  - Leyenburg Hospital; Pulmonology, The Hague
- College of Medicine & Sciences, Sultan Qaboos University Hospital, Muscat, Oman
- Slovakia (4):
  - Fnsp Fdr Banska Bystrica; Dep of Pneumology&Ftizeology, Banská Bystrica
  - FNsP Bratislava, Nemocnica Ruzinov, Bratislava
  - Vychodoslovensky onkologicky ustav, Košice
  - Inst. of Tb & Respiratory Diseases; Dep. of Oncology, Nitra
- Spain (8):
  - Hospital de Cruces; Servicio de Oncologia, Barakaldo, Vizcaya
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Centro Oncologico MD Anderson International Espana, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Tawam Hospital; Medical Oncology Department, Al Ain City, United Arab Emirates

REFERENCES:
- [Derived] Gridelli C, de Castro Carpeno J, Dingemans AC, Griesinger F, Grossi F, Langer C, Ohe Y, Syrigos K, Thatcher N, Das-Gupta A, Truman M, Donica M, Smoljanovic V, Bennouna J. Safety and Efficacy of Bevacizumab Plus Standard-of-Care Treatment Beyond Disease Progression in Patients With Advanced Non-Small Cell Lung Cancer: The AvaALL Randomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):e183486. doi: 10.1001/jamaoncol.2018.3486. Epub 2018 Dec 13. PMID 30177994
- [Derived] Takeda M, Yamanaka T, Seto T, Hayashi H, Azuma K, Okada M, Sugawara S, Daga H, Hirashima T, Yonesaka K, Urata Y, Murakami H, Saito H, Kubo A, Sawa T, Miyahara E, Nogami N, Nakagawa K, Nakanishi Y, Okamoto I. Bevacizumab beyond disease progression after first-line treatment with bevacizumab plus chemotherapy in advanced nonsquamous non-small cell lung cancer (West Japan Oncology Group 5910L): An open-label, randomized, phase 2 trial. Cancer. 2016 Apr 1;122(7):1050-9. doi: 10.1002/cncr.29893. Epub 2016 Feb 1. PMID 26828788
- [Derived] Gridelli C, Bennouna J, de Castro J, Dingemans AM, Griesinger F, Grossi F, Rossi A, Thatcher N, Wong EK, Langer C. Randomized phase IIIb trial evaluating the continuation of bevacizumab beyond disease progression in patients with advanced non-squamous non-small-cell lung cancer after first-line treatment with bevacizumab plus platinum-based chemotherapy: treatment rationale and protocol dynamics of the AvaALL (MO22097) trial. Clin Lung Cancer. 2011 Nov;12(6):407-11. doi: 10.1016/j.cllc.2011.05.002. Epub 2011 Jun 25. PMID 21705281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 3b study was conducted across 16 different countries and enrolled 485 participants. Participants were 18 years or older and had locally recurrent or metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC)
Pre-assignment Details: A total of 485 participants were enrolled and randomized into the study. Of these, 475 participants were treated; 243 participants received bevacizumab plus standard of care (SoC) and 232 participants received SoC alone. The study was terminated 60 months after study start, as per protocol, but was not ended prematurely.
Groups:
- Bevacizumab + Standard of Care: Participants received bevacizumab on Day 1 of every 21-days cycle along with standard of care, until the occurrence of an unacceptable toxicity or withdrawal of consent (whichever occurs first).
- Standard of Care: Participants received investigator's choice of standard of care (Erlotinib or Docetaxel or Pemetrexed) according to local practice until the occurrence of an unacceptable toxicity or withdrawal of consent (whichever occurs first).
Period: Overall Study
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Started | 245 | 240
Treated Participants | 243 | 232
Completed | 0 | 0
Not Completed | 245 | 240
Not completed — Withdrawal by Subject | 15 | 17
Not completed — Trial termination by the Sponsor | 28 | 19
Not completed — Lost to Follow-up | 5 | 7
Not completed — Death | 190 | 187
Not completed — Physician Decision | 2 | 3
Not completed — Reason unknown | 0 | 2
Not completed — Never Started | 5 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 245 | 240 | 485
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (9.61) [26 to 84] | 61.8 (9.29) [35 to 82] | 61.6 (9.44) [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 102 | 192
  Male | 155 | 138 | 293

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of randomization at first progression of disease to the date of death, regardless of the cause of death.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Months | 11.86 [10.22 to 13.67] | 10.22 [8.61 to 11.93]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; The stratification factors for Log-Rank test and Hazard Ratio (HR) are the type of planned 2nd-line SoC treatment, the number of cycles of bevacizumab maintenance treatment prior to first PD and smoking status; Test type: Superiority or Other; p = 0.1044, Stratified Log-Rank test; Stratified Hazard Ratio = 0.84, 90% CI 2-sided [0.71 to 1.00]

2. Secondary Outcome: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was defined as the time from start of treatment to the first event of death or PD. Tumor response was assessed by the IRF according to RECIST v1.1. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PFS2 is defined as the time between randomization at PD1 and the date of PD2 or death, whichever occurs first. PFS3 is defined as the time between PD2 and the date of PD3 or death, whichever occurs first.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Months
  PFS 2 | 5.45 [4.21 to 5.68] | 3.98 [3.38 to 4.30]
  PFS 3 | 4.01 [2.86 to 4.47] | 2.60 [2.33 to 2.92]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; PFS 2: The stratification factors for Log-Rank test are the type of planned 2nd-line SoC treatment, the number of cycles of bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0573, Stratified Log-Rank test; Stratified Hazard Ratio = 0.83, 90% CI 2-sided [0.70 to 0.98]
Statistical Analysis 2: Comparison: Bevacizumab + Standard of Care vs Standard of Care; PFS 3: The stratification factors for Log-Rank test are the type of planned 2nd-line SoC treatment, the number of cycles of bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0045, Stratified Log-Rank test; Stratified Hazard Ratio = 0.63, 90% CI 2-sided [0.49 to 0.83]

3. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST v1.1
Description: The objective response is defined as complete response (CR) or partial response (PR) assessed according to the RECIST v.1.1 criteria with baseline tumour assessment as the reference. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Percentage of Participants | 8.6 [5.86 to 12.21] | 6.3 [3.91 to 9.50]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; The stratification factors for Cochran-Mantel-Haenszel test are the type of planned 2nd-line SoC treatment, the number of cycles of Bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0810, Stratified Cochran-Mantel-Haenszel test; Estimated difference in response rate = 0.0237, 90% CI 2-sided [-0.0156 to 0.0630]

4. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST v1.1
Description: The disease control rate is defined as CR or PR or stable disease (SD) assessed according to the RECIST v.1.1 criteria with baseline tumour assessment as the reference. SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment started for target lesions and the persistence of 1 or more non-target lesions.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Percentage of Participants | 80.2 [75.57 to 84.36] | 77.0 [72.06 to 81.41]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0218, Stratified Cochran-Mantel-Haenszel test; Estimated difference in Disease Control = 0.0326, 90% CI 2-sided [-0.0288 to 0.0940]

5. Secondary Outcome: Duration of Response (DoR) According to RECIST v1.1
Description: Duration of response is defined as the time that measurement criteria are met for objective response (CR/PR) (whichever status is recorded first) until the first date of progression or death is documented. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than < 10 mm. PR was defined as greater than or equal to ≥30 % decrease in sum of longest diameter of target lesions in reference to baseline sum longest diameter.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Months | 7.46 [5.39 to 8.54] | 6.24 [3.52 to 6.83]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; The stratification factors for Log-Rank test are the type of planned 2nd-line SoC treatment, the number of cycles of Bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0600, Stratified Log-Rank test; Stratified Hazard Ratio = 0.29, 90% CI 2-sided [0.09 to 0.90]

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: The safety population included all participants who had received at least one dose of any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 243 | 232
Percentage of Participants
  AEs | 97.5 | 96.1
  SAEs | 51.9 | 37.1

7. Secondary Outcome: Time to Progression (TTP) According to RECIST v1.1
Description: The time to progression was defined as the time from baseline until disease progression as determined by the RECIST v1.1. TTP2 is defined as the interval between the day of randomization at PD1 and PD2. TTP3 is defined as the interval between the day of PD2 and PD3. PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Population: Intent to treat population included all randomized participants.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Months
  TTP2 | 5.55 [4.86 to 6.18] | 4.21 [3.75 to 5.06]
  TTP3 | 4.07 [3.25 to 4.63] | 2.73 [2.37 to 3.06]
Statistical Analysis 1: Comparison: Bevacizumab + Standard of Care vs Standard of Care; TTP2: The stratification factors for Log-Rank test are the type of planned 2nd-line SoC treatment, the number of cycles of Bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0311, Stratified Log-Rank test; Stratified Hazard Ratio = 0.79, 90% CI 2-sided [0.65 to 0.95]
Statistical Analysis 2: Comparison: Bevacizumab + Standard of Care vs Standard of Care; TTP3: The stratification factors for Log-Rank test are the type of planned 2nd-line SoC treatment, the number of cycles of Bevacizumab maintenance treatment prior to PD1 and the smoking status; Test type: Superiority or Other; p = 0.0326, Stratified Log-Rank test; Stratified Hazard Ratio = 0.69, 90% CI 2-sided [0.52 to 0.92]

8. Secondary Outcome: Percentage of Participants Who Are Alive at Month 6, 12, and 18
Description: Percentage of participants who were alive at Month 6, 12 and 18 were reported.
Time Frame: Month 6, 12, 18
Population: Intent to treat population included all randomized participants.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Number analyzed (Participants) | 245 | 240
Percentage of Participants
  Month 6 | 0.8 [0.73 to 0.82] | 0.7 [0.62 to 0.72]
  Month 12 | 0.5 [0.44 to 0.54] | 0.4 [0.39 to 0.50]
  Month 18 | 0.4 [0.31 to 0.41] | 0.3 [0.25 to 0.36]

ADVERSE EVENTS:
Time Frame: Up to data cut-off date 24 June 2016 (approximately 5 years)
Description: The safety population included all participants who had received at least one dose of any study drug.
Arm/Group | Bevacizumab + Standard of Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 126/243 | 86/232
Other Adverse Events (participants affected / at risk) | 226/243 | 215/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Standard of Care (N=243) | Standard of Care (N=232)
Anaemia (Blood and lymphatic system disorders) | 2 | 6
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 12 | 9
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 6
Pure White Cell Aplasia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 1
Cardiac Failure (Cardiac disorders) | 1 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Tracheo-oesophageal Fistula (Congenital, familial and genetic disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 2 | 0
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 4 | 0
Death (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 2
General Physical Health Deterioration (General disorders) | 1 | 2
Malaise (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 3 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Performance Status Decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 1
Sudden Death (General disorders) | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Anal Abcess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0
Device related Infection (Infections and infestations) | 1 | 1
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Febrile Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Genital Herpes Simplex (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lung Abcess (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 3 | 1
Periorbital Abcess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 13 | 19
Post Procedural Infection (Infections and infestations) | 1 | 0
Psoas Abcess (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 6 | 1
Respiratory tract Infection Bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic Shock (Infections and infestations) | 0 | 1
Subcutaneous Abcess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Arterial Injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 3 | 0
Liver Function Test Increased (Investigations) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Tetany (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervetebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Parapalegia (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Apathy (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 2
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Prerenal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Tubular Disorder (Renal and urinary disorders) | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organizing Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Osteosynthesis (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Peripheral Embolism (Vascular disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Standard of Care (N=243) | Standard of Care (N=232)
Anaemia (Blood and lymphatic system disorders) | 54 | 69
Leukopenia (Blood and lymphatic system disorders) | 16 | 10
Neutropenia (Blood and lymphatic system disorders) | 39 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 9
Lacrimation Increased (Eye disorders) | 18 | 12
Abdominal Pain (Gastrointestinal disorders) | 16 | 13
Abdominal Pain Upper (Gastrointestinal disorders) | 25 | 14
Constipation (Gastrointestinal disorders) | 64 | 49
Diarrhoea (Gastrointestinal disorders) | 90 | 72
Nausea (Gastrointestinal disorders) | 84 | 61
Stomatitis (Gastrointestinal disorders) | 39 | 26
Vomiting (Gastrointestinal disorders) | 51 | 40
Asthenia (General disorders) | 68 | 61
Chest Pain (General disorders) | 26 | 16
Fatigue (General disorders) | 71 | 73
Malaise (General disorders) | 24 | 14
Mucosal Inflammation (General disorders) | 49 | 22
Oedema Peripheral (General disorders) | 34 | 32
Pain (General disorders) | 10 | 13
Pyrexia (General disorders) | 46 | 35
Bronchitis (Infections and infestations) | 23 | 12
Conjunctivitis (Infections and infestations) | 16 | 13
Pneumonia (Infections and infestations) | 9 | 12
Respiratory Tract Infection (Infections and infestations) | 13 | 9
Urinary Tract Infection (Infections and infestations) | 16 | 10
Blood Creatinine Increased (Investigations) | 13 | 4
Weight Decreased (Investigations) | 42 | 24
Decreased Appetite (Metabolism and nutrition disorders) | 83 | 59
Dehydration (Metabolism and nutrition disorders) | 13 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 28 | 31
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 13 | 8
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 22 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 18
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 17 | 16
Dizziness (Nervous system disorders) | 20 | 13
Dysgeusia (Nervous system disorders) | 29 | 16
Headache (Nervous system disorders) | 39 | 23
Neuropathy Peripheral (Nervous system disorders) | 20 | 16
Paraesthesia (Nervous system disorders) | 15 | 8
Anxiety (Psychiatric disorders) | 11 | 12
Insomnia (Psychiatric disorders) | 14 | 15
Proteinuria (Renal and urinary disorders) | 51 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 40
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 56
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 | 20
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 55 | 41
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 15 | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 29 | 22
Erythema (Skin and subcutaneous tissue disorders) | 11 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 14
Rash (Skin and subcutaneous tissue disorders) | 49 | 46
Hypertension (Vascular disorders) | 52 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.